CLINICAL TRIAL: NCT02670460
Title: Percutaneous Temporary Placement of a Phrenic Nerve Stimulator for Diaphragm Pacing, a First in Human Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lungpacer Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TPR-0046 and CLN-0005
Record Dates: First submitted 2016-01-27; First posted 2016-02-01 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Ventilator Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temporary diaphragmatic pacing (Experimental): There is no comparator for this study. Single site and all patients are in the treatment allocated group of temporary diaphragmatic pacing with the LIVE Catheter which is inserted via the left subclavian vein.
  Interventions: Device: LIVE Catheter

INTERVENTIONS:
Device: LIVE Catheter — Placement of a temporary LIVE Catheter central venous pacing device in the left subclavian vein to pace the phrenic nerves and allow recruitment of the diaphragm muscle.

SUMMARY:
Study conducted to confirm phrenic nerve stimulation using the Lungpacer LIVE Catheter, confirm capture of the diaphragm and confirm that the diaphragm can be paced in synchrony with mechanical ventilator breaths.

DETAILED DESCRIPTION:
This study is being conducted to determine if in an anaesthetized (sedated, intubated and mechanically ventilated) subject the LIVE Catheter can be inserted percutaneously and activated via the electrical stimulator to stimulate the left and right phrenic nerves causing the diaphragm to contract in synchrony with mechanical ventilator breaths via phrenic nerve stimulation from a transvenously delivered electrical current.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent or whose legally authorized representative is able and willing to give informed consent.
* Able to undergo general anaesthesia (sedation, intubation and mechanical ventilation)
* Susceptible indication for atrial septal defect closure

Exclusion Criteria:

* Subject has an EF of < 30%
* Subject has a co-morbid illness or life expectancy < 2 years
* Subject has experienced an AMI within 72 hours prior to this procedure
* Subject is contraindicated for or unwilling to take aspirin or anticoagulants
* Subject is in cardiogenic shock
* Subject has other cardiovascular disease requiring open heart surgery
* Subject is known to have a demonstrated intra cardiac thrombus on echocardiography
* Subject has been treated with paralytic medications within 72 hours prior to procedure
* Subject has significant thoracic abnormalities such that placement of a left subclavian line would be difficult
* Inability to cannulate the left subclavian vein (post-consent exclusion)
* Subject has a known or suspected phrenic nerve paralysis
* Subject has co-existing temporary or implanted cardiac electrical devices such as a pacemaker or defibrillator
* Subject has an active systemic infection or local infection at or around the insertion site
* Subject is known or suspected to be pregnant or is lactating
* Subject will be unavailable for, or is unwilling to comply with, follow up requirements of the protocol
* Subject is currently enrolled in any other study of an investigational drug or device who has received treatment under that protocol with the investigational product during the 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Successful insertion of the LIVE Catheter into the left subclavian vien | at time of procedure
  Confirmation by cinefluoroscopy of the insertion of the LIVE Catheter into the Left subclavian vein with the tip located in the superior vena cava
Absence of device related or procedure related adverse events | up to 48 hours or at time of discharge whichever comes first
  Assess subject AE status out to 48 hours post procedure

SECONDARY OUTCOMES:
Phrenic nerve stimulation in synchrony with MV breaths | No more than 90 minutes procedure duration
  Phrenic nerve stimulation in synchrony with MV breaths as defined by contraction of the diaphragm upon energy delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Reynolds, MD, Study Director — Lungpacer Medical
Locations (1):
- Italian Hospital, Asunción, Casa Zanotti, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided
Discussing a publication for FIH

REFERENCES:
- [Background] Penuelas O, Frutos-Vivar F, Fernandez C, Anzueto A, Epstein SK, Apezteguia C, Gonzalez M, Nin N, Raymondos K, Tomicic V, Desmery P, Arabi Y, Pelosi P, Kuiper M, Jibaja M, Matamis D, Ferguson ND, Esteban A; Ventila Group. Characteristics and outcomes of ventilated patients according to time to liberation from mechanical ventilation. Am J Respir Crit Care Med. 2011 Aug 15;184(4):430-7. doi: 10.1164/rccm.201011-1887OC. PMID 21616997
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Supinski GS, Callahan LA. Diaphragm weakness in mechanically ventilated critically ill patients. Crit Care. 2013 Jun 20;17(3):R120. doi: 10.1186/cc12792. PMID 23786764
- [Background] Gayan-Ramirez G. Ventilator-induced diaphragm dysfunction: time for (contr)action! Eur Respir J. 2013 Jul;42(1):12-5. doi: 10.1183/09031936.00076513. No abstract available. PMID 23813310